CLINICAL TRIAL: NCT01629849
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 1021958 Tablets in Otherwise Healthy Controlled Asthmatic Subjects (Phase I, Randomised, Placebo-controlled, Double-blind Within Dose Groups)
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 1021958 in Otherwise Healthy Controlled Asthmatic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1310.2; 2012-000926-23 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-06-21; First posted 2012-06-28 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Healthy; Asthma
MeSH Terms: conditions — Asthma

ARMS (4):
- BI 1021958 qd (Experimental): Multiple rising dose
  Interventions: Drug: BI 1021958 qd
- Placebo to BI 1021958 qd (Placebo Comparator): Matching placebo as tablets
  Interventions: Drug: Placebo to BI 1021958 qd
- BI 1021958 bid (Experimental): Multiple rising dose
  Interventions: Drug: BI 1021958 bid
- Placebo to BI 1021958 bid (Placebo Comparator): Matching palcebo as tablet
  Interventions: Drug: Placebo to BI 1021958 bid

INTERVENTIONS:
Drug: Placebo to BI 1021958 qd — tablet
  Arms: Placebo to BI 1021958 qd
Drug: BI 1021958 bid — tablets
  Arms: BI 1021958 bid
Drug: Placebo to BI 1021958 bid — tablets
  Arms: Placebo to BI 1021958 bid
Drug: BI 1021958 qd — tablet
  Arms: BI 1021958 qd

SUMMARY:
To investigate safety, tolerability, pharmacokinetics including posology, and pharmacodynamics of multiple rising doses of BI 1021958 in otherwise healthy mild asthmatic subjects

ELIGIBILITY:
Inclusion criteria:

1. Healthy male and female subjects ofn non child-bearing potential

Exclusion criteria:

1. Any relevant deviation from healthy conditions except mild controlled asthma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with drug-related adverse events | up to day 22

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte in plasma) | up to 481:30 h
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | up to 481:30 h
AUCt,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval t after administration of the first dose) | up to 481:30 h
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point within the first dosing interval) | up to 481:30 h
AUC0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 481:30 h
Cpre,N (predose concentration of the analyte in plasma immediately before administration of the Nth dose after N-1 doses were administered | up to 481:30 h
terminal rate constant in plasma | up to 481:30 h
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 481:30 h
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval t) | up to 481:30 h
tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) | up to 481:30 h
Cmin,ss (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval t) | up to 481:30 h
AUCt,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval t) | up to 481:30 h
terminal rate constant in plasma at steady state | up to 481:30 h
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | up to 481:30 h
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | up to 481:30 h
CL/F,ss (apparent clearance of the analyte in the plasma at steady state following extravascular multiple dose administration) | up to 481:30 h
Vz/F,ss (apparent volume of distribution during the terminal phase at steady state following extravascular administration) | up to 481:30 h
Cavg (average concentration) | up to 481:30 h
PTF (peak trough fluctuation) | up to 481:30 h

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1310.2.1 Boehringer Ingelheim Investigational Site, Gauting, Germany